CLINICAL TRIAL: NCT01640535
Title: Efficacy and Safety of Concomitant Montelukast Sodium and Levocetirizine Dihydrochloride in Perennial Allergic Rhinitis (PAR) Patients : A Randomized, Double-blind, Active-controlled, Multicenter Phase 3 Clinical Trial
Brief Title: Efficacy and Safety of Concomitant Montelukast Sodium and Levocetirizine Dihydrochloride in Perennial Allergic Rhinitis (PAR) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM-MOLZ-301
Record Dates: First submitted 2012-07-10; First posted 2012-07-13 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Perennial Allergic Rhinitis
Keywords: PAR
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — montelukast; levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test arm (Experimental): Montelukast sodium 10 mg + Levocetirizine dihydrochloride 5 mg
  Interventions: Drug: Montelukast + Levocetirizine
- Comparator arm I (Active Comparator): Matching placebo of Montelukast sodium 10mg + Levocetirizine dihydrochloride 5 mg
  Interventions: Drug: Levocetirizine
- Comparator arm II (Active Comparator): Montelukast sodium 10mg + matching placebo of Levocetirizine dihydrochloride 5mg
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast + Levocetirizine — Tablet, Montelukast sodium 10 mg + Levocetirizine dihydrochloride 5 mg, Once daily (before bedtime)
  Other Names: Singulair Tablet, Xyzal Tablet
  Arms: Test arm
Drug: Levocetirizine — Tablet, Matching placebo of Montelukast sodium 10 mg + Levocetirizine dihydrochloride 5 mg, Once daily (before bedtime)
  Other Names: Xyzal Tablet
  Arms: Comparator arm I
Drug: Montelukast — Tablet, Montelukast sodium 10 mg + matching placebo of Levocetirizine dihydrochloride 5 mg, Once daily (before bedtime)
  Other Names: Singulair Tablet
  Arms: Comparator arm II

SUMMARY:
The purpose of this study is to demonstrate that the efficacy of Concomitant Montelukast Sodium and Levocetirizine Dihydrochloride is superior to that of Levocetirizine and Montelukast monotherapies and to compare the safety and tolerability of Concomitant Montelukast Sodium and Levocetirizine Dihydrochloride to those of Levocetirizine and Montelukast monotherapies in Perennial Allergic Rhinitis (PAR) patients.

DETAILED DESCRIPTION:
randomized, double-blind, active-controlled, multicenter, phase 3 trial

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 2 years history of PAR prior to the study
* Positive results of skin prick test
* Patients who provided a signed written informed consent form
* Patients who are able and willing to complete subject diaries
* Patients who agree to maintain consistency in their surroundings throughout the study period
* At Visit, 2 patients whose symptom scores recorded in the subject diary meet all of the followings during the last one week of baseline period A.Daily mean of 6 points or above for Daytime Nasal Symptom Score (maximum 12 points) B.Daily mean of 1.8 points or above for Daytime Nasal Obstruction Symptom Score (maximum 3 points)

Exclusion Criteria:

* Patients also with non-allergic rhinitis with different causes.
* Patients with severe asthma who meet the followings.
* Presence of nasal polyps or any clinically important nasal anomaly.
* History of acute • chronic sinusitis within 30 days of Visit 1
* History of intranasal / eye surgeries within 3 months of Visit 1
* Initiation of immunotherapy or dose modification within 1 month prior to Visit 1
* Upper respiratory infections including cold and systemic infections within 3 weeks of Visit 1.
* Chronic use of tricyclic antidepressants, beta agonists, bronchodilators, etc. that may affect the efficacy of study drug
* At Visit 2, patients who recorded Daytime Nasal Symptom Scores for fewer than 4 days in the subject diary during the last one week of baseline period

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Mean Daytime Nasal Symptom Score | 4 weeks
  Change in Mean Daytime Nasal Symptom Score from baseline at Weeks 3-4(2 weeks) of treatment

SECONDARY OUTCOMES:
Change in Mean Nighttime Nasal Symptom from baseline at Weeks 1-2 (2 weeks) and Weeks 3-4 (2 weeks) of treatment | 4 weeks
  Change in Mean Nighttime Nasal Symptom from baseline at Weeks 1-2 (2 weeks) and Weeks 3-4 (2 weeks) of treatment
Mean Composite Symptom Score | 4 weeks
  Change in Mean Composite Symptom Score from baseline at Weeks 1-2 (2 weeks) and Weeks 3-4 (2 weeks) of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyungmi PARK, PhD, Study Director — Hanmi Pharmaceutical Company Limited
Locations (1):
- Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do, South Korea